CLINICAL TRIAL: NCT00017264
Title: A Phase I Evaluation of the Safety and Pharmacokinetics of ABT-627 in Adults With Recurrent Malignant Gliomas
Brief Title: Atrasentan in Treating Patients With Progressive or Recurrent Malignant Glioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068668; NABTT-2008; JHOC-NABTT-2008
Record Dates: First submitted 2001-06-06; First posted 2003-01-27 (Estimated); Last update posted 2009-01-13 (Estimated); Status verified 2004-08

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent adult brain tumor; adult glioblastoma; adult anaplastic astrocytoma; adult anaplastic oligodendroglioma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Glioblastoma; Astrocytoma; Oligodendroglioma; Gliosarcoma | interventions — Atrasentan

INTERVENTIONS:
Drug: atrasentan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of atrasentan in treating patients who have progressive or recurrent malignant glioma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of atrasentan in patients with progressive or recurrent malignant glioma.
* Describe the pharmacokinetics of this drug in these patients.
* Assess preliminary evidence of therapeutic activity of this drug in these patients.

OUTLINE: This is a dose-escalation, multicenter study.

Patients receive oral atrasentan once daily. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 2-10 patients receive escalating doses of atrasentan until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 1 patient experiences dose-limiting toxicity.

Patients are followed every 2 months.

PROJECTED ACCRUAL: Approximately 35 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignant glioma

  * Anaplastic astrocytoma
  * Anaplastic oligodendroglioma
  * Glioblastoma multiforme
* Progressive or recurrent after prior radiotherapy with or without chemotherapy

  * Prior low-grade glioma that has progressed to high-grade after therapy allowed
* Measurable disease by MRI or CT scan

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 mg/dL
* Transaminases no greater than 4 times upper limit of normal
* Hepatitis A, B, and C negative

Renal:

* Creatinine no greater than 1.7 mg/dL

Cardiovascular:

* No New York Heart Association class II, III, or IV cardiac disease

Other:

* HIV negative
* Mini mental score at least 15
* No other malignancy within the past 5 years except curatively treated carcinoma in situ or basal cell skin cancer
* No serious concurrent infection
* No other concurrent medical illness that would preclude study entry
* No alcoholism or drug addiction within the past 6 months
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent anticancer immunotherapy

Chemotherapy:

* See Disease Characteristics
* At least 3 weeks since prior chemotherapy (6 weeks for nitrosoureas) and recovered
* No more than 1 prior chemotherapy regimen
* No prior or concurrent polifeprosan 20 with carmustine implant (Gliadel wafer)
* No prior atrasentan
* No other concurrent anticancer chemotherapy

Endocrine therapy:

* No concurrent anticancer hormonal therapy

Radiotherapy:

* See Disease Characteristics
* At least 3 months since prior radiotherapy and recovered
* No concurrent anticancer radiotherapy

Surgery:

* No concurrent anticancer surgery

Other:

* Recovered from prior therapy
* No more than 1 prior treatment regimen
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-06

CONTACTS AND LOCATIONS:
Overall Officials: Surasak Phuphanich, MD, FAAN, Study Chair — Emory University
Locations (10):
- United States (10):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Abramson Cancer Center at University of Pennsylvania Medical Center, Philadelphia, Pennsylvania
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas

REFERENCES:
- [Result] Phuphanich S, Carson KA, Grossman SA, Lesser G, Olson J, Mikkelsen T, Desideri S, Fisher JD; New Approaches to Brain Tumor Therapy (NABTT) CNS Consortium. Phase I safety study of escalating doses of atrasentan in adults with recurrent malignant glioma. Neuro Oncol. 2008 Aug;10(4):617-23. doi: 10.1215/15228517-2008-013. Epub 2008 May 13. PMID 18477765